CLINICAL TRIAL: NCT02809456
Title: Mitigation of Radiation Pneumonitis, Fibrosis and Heart Toxicity With Nicorandil in Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Szu-Yuan Wu, Department of Radiation Oncology, Taipei Medical University WanFang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N201508038
Record Dates: First submitted 2016-06-09; First posted 2016-06-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis | interventions — Nicorandil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil (Experimental): Beginning 4-6 weeks during radiation therapy, patients receive nicorandil is given during radiotherapy interval, 5mg each time, 3 times daily oral. Treatment repeats after completion of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nicorandil
- observation (Active Comparator): regular radiotherapy as our protocol
  Interventions: Drug: Nicorandil

INTERVENTIONS:
Drug: Nicorandil — oral intake
  Other Names: Ikorel; Angedil; Dancor; Nikoran,PCA; Aprior; Nitorubin; Sigmart

SUMMARY:
This project will test the effect of nicorandil to mitigate the lung damage that can occur as a side effect of radiation therapy for lung cancer. Thousands of veterans develop lung cancer every year, and are treated by radiation therapy. Studies of lung radiation injury in laboratory animals show that with nicorandil, investigators can significantly reduce the severity of lung fibrosis and heart toxicity.1,2 Nicorandil is FDA approved and in common use for treatment of angina. These studies will advance that work to human use. Successful mitigation of lung radiation damage and heart toxicity will improve the quality of life in veterans and non-veterans who are treated for lung cancer by radiation, and may also improve cure rates of radiation therapy for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-proven NSCLC; mixed histology with small cell lung carcinoma (SCLC) component not allowed
2. Patients with stage II - IV NSCLC who received at least 54 Gy of total planned thoracic radiation dose will be eligible; patients must have received at least one cycle of chemotherapy concurrently during the course of thoracic radiation; regimens allowed are platinum combinations with either etoposide or a taxane regardless of histology subtype; platinum with pemetrexed for patients with nonsquamous NSCLC only; patients with oligometastatic stage IV cancer are eligible if they have received only one line of systemic therapy for their stage IV cancer prior to the concurrent chemoradiation phase
3. Patient must have had a CR/PR/SD, 4-6 weeks after completing last fraction of chemotherapy / radiation therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance score 0-2 at the time of randomization
5. Absolute neutrophil count (ANC) >= 1,500/uL
6. Platelet count >= 100,000/uL
7. Hemoglobin >= 9 g/dL
8. Total bilirubin =< 1.5 times upper limit of normal (ULN) OR direct bilirubin normal (per institute standards)
9. Aspartate aminotransferase (AST) =< 1.5 x ULN; alanine aminotransferase (ALT) and AST =< 3 x ULN is acceptable if there is liver metastasis
10. Fertile patients must use adequate contraception

Exclusion Criteria:

1. Whole-brain radiotherapy (WBRT) < 14 days from the anticipated start of nicorandil/placebo administration
2. Unable to start nicorandil/placebo treatment between 4 - 6 weeks after completing the last dose of thoracic radiation
3. Active untreated brain or leptomeningeal metastases; in patients with treated central nervous system (CNS) metastases, eligible if symptoms controlled for at least 4 weeks; dexamethasone allowed if total daily dose does not exceed 2 mg
4. Major injuries or surgery (e.g., craniotomy) < 28 days from the start of nicorandil/placebo administration; wound should be healed prior to starting therapy
5. Second malignancies are allowed as long as the disease does not require active treatment with concomitant systemic cytotoxic chemotherapy, investigational or biologic therapy (e.g., anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA4] or human epidermal growth factor receptor 2 [HER2] monoclonal antibodies); hormone-related therapies (e.g., gonadotrophin releasing hormone (LHRH) agonists, tamoxifen, etc.) are allowed
6. Concurrent uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would increase the risk associated with study participation and/or limit compliance with study requirements
7. Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher proteinuria
8. Systemic therapy or investigational agent administered < 28 days prior to treatment with nicorandil
9. Pregnancy or breast feeding; female patients with child-bearing potential must have a negative pregnancy test (beta-human chorionic gonadotropin [B-HCG] test in urine or serum) prior to commencing study treatment
10. Creatinine > 1.5 x ULN or creatinine clearance levels (CrCL) < 45 mL/min
11. Centrally located tumors with radiographic evidence (computed tomography [CT] or magnetic resonance imaging [MRI]) of local invasion of major blood vessels
12. acute myocardial infarction within 2 weeks before percutaneous coronary intervention
13. contraindications to treatment with nicorandil (allergy, glaucoma, digestive ulcer, is currently taking phosphodiesterase-5 inhibitor)
14. bypass restenosis
15. PCI history
16. hypotension
17. impaired liver function
18. renal insufficiency requiring hemodialysis
19. pregnancy
20. connective tissue disease
21. life expectancy ≤ 12 months
22. left main coronary artery disease
23. bypass graft lesion and lesions unsuitable for OCT
24. unwillingness or inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The rate of symptomatic radiation pneumonitis in patients with unresectable Stage II/III/ oligometastatic IV non-small cell lung carcinoma (NSCLC) who completed chemoradiation followed by nicorandil or not | Up to 2.5 years post-treatment

SECONDARY OUTCOMES:
The quality of life (QOL) questionnaire | Baseline up to 2.5 years post-treatment
Biomarker analysis such as TGF-β, Serum surfactant proteins-A & -D, MMP1 and MMP7 | Up to 97 days post-treatment
The overall survival in patients who received nicorandil versus observation | Up to 2.5 years post-treatment
Radiation pneumonitis (RP) score in patients who received nicorandil versus observation | Baseline up to 2.5 years post-treatment
The composite index (based on PFT, RP score and QOL) at the end of active treatment and 6 months after completion of treatment between patients who received nicorandil versus observation. | Baseline up to 2.5 years post-treatment
Responses rates | Up to 2.5 years post-treatment

IPD SHARING:
Plan to Share IPD: Undecided